CLINICAL TRIAL: NCT05527509
Title: Risk and Resiliency Factors in the RCMP: A Prospective Investigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Royal Canadian Mounted Police (Unknown); Government of Canada (Other Government); Ministry of Public Safety and Emergency Preparedness (Unknown); Canadian Institute for Public Safety Research and Treatment (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-055
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Posttraumatic Stress Disorder; Major Depressive Disorder; Panic Disorder; Generalized Anxiety Disorder; Trauma; Traumatic Stress Disorder; Trauma and Stress Related Disorders; Vicarious Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Panic Disorder; Generalized Anxiety Disorder; Wounds and Injuries; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders; Compassion Fatigue

STUDY DESIGN:
Intervention Model Description: The RCMP Study necessarily uses a longitudinal prospective sequential experimental cohort design to create a clustered randomized trial that engages individual participants for 5.5 years. The structure of the Cadet Training Program does not allow for randomizing individual participants or individual groups of participants; nevertheless, meta-analytic evidence suggests that results from studies using this design and results from true randomized controlled trials do not typically differ meaningfully or statistically significantly, and both methods produce comparable groups at baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Training Condition (STC) (Active Comparator): The STC has received the "standard" RCMP Depot Division ("Depot") Cadet Training Program as has been provided to cadets prior to June 2022. The STC and the ATC will complete the same standardized self-report assessments, clinical interview assessments, and biometric assessments, and receive the same feedback and reporting based on those assessments.
  Interventions: Behavioral: Active Monitoring
- Augmented Training Condition (ATC) (Experimental): The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) is an evidence-based cognitive-behavioral intervention designed to cultivate constructive approach-oriented emotional engagement. The 13-week Emotional Resilience Training (ERST) is an adaptation of the UP designed for use as a proactive training course. The ERST frames emotional experiences as natural responses to threat, rather than pathological occurrences to avoid; as such, the ERST is well-suited for mitigating health challenges and the skills may also help PSP to support persons in distress, including other PSP and the community members they all serve. The ERST training materials include an instructor guide, didactic PowerPoints, and a trainee workbook. The ERST was designed for seamless integration with the Cadet Training Program, effective June 2022, which is what creates the augmented training arm (i.e., the ATC).
  Interventions: Behavioral: Emotional Resilience Skills Training (ERST)

INTERVENTIONS:
Behavioral: Emotional Resilience Skills Training (ERST) — The ERST training is designed as a "train the trainer" model. Sauer-Zavala, a co-developer of the UP, personally trained a group of RCMP trainers during a week-long interactive workshop. The trainers continue to have access to Sauer-Zavala for optional follow-up consultation and support related to delivery of the ERST training for questions or to address any issues that arise during training. Having consultation and support available for the trainers should help to offset concerns raised about ensuring training fidelity subsequent to other mental health programs. Participants have ongoing access to ERST to support skill retention after training is completed, which should help to offset previous indications of problems with skill development for mental health programs.
  Other Names: Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP)
  Arms: Augmented Training Condition (ATC)
Behavioral: Active Monitoring — Participants in the STC will be assessed for at least 66 months, via full assessments (i.e., self-report surveys, clinical interviews), monthly assessments (i.e., ~20 minute self-report surveys), daily assessments (i.e., ~1 minute self-report surveys), and biometric assessments. The self-monitoring and feedback should be inherently beneficial and should facilitate earlier access to evidence-based care, which is why the STC is considered an active comparator.
  Arms: Standard Training Condition (STC)

SUMMARY:
The Royal Canadian Mounted Police (RCMP), like all public safety personnel (PSP), are frequently exposed to potentially psychologically traumatic events that contribute to posttraumatic stress injuries (PTSI). Addressing PTSI is impeded by the limited available research. The RCMP are working to build evidence-based solutions to PTSI and other mental health challenges facing their members, which by extension will help all PSP, as part of the Canadian Government Federal Framework on Posttraumatic Stress Disorder. A key element is the "Longitudinal Study of Operational Stress Injuries / Étude longitudinale sur les traumatismes liés au stress opérationnel", a study which has been renamed "Risk and Resiliency Factors in the RCMP: A Prospective Investigation", and is referred to as the "RCMP Study" for short. The RCMP Study has been detailed online (www.rcmpstudy.ca) and in a recently published peer-reviewed protocol paper, "The Royal Canadian Mounted Police (RCMP) Study: protocol for a prospective investigation of mental health risk and resilience factors" (https://doi.org/10.24095/hpcdp.42.8.02). The RCMP Study, part of the concerted efforts by the RCMP to reduce PTSI by improving access to evidence-based assessments, treatments, and training as well as participant recruitment and RCMP Study developments to date. The RCMP Study has been designed to (1) develop, deploy and assess the impact of a system for ongoing annual, monthly and daily evidence-based assessments; (2) evaluate associations between demographic variables and PTSI; (3) longitudinally assess individual differences associated with PTSI; (4) augment the RCMP Cadet Training Program with skills to proactively mitigate PTSI; and (5) assess the impact of the augmented training condition (ATC) versus the standard training condition (STC). Participants in the STC (n = 480) and ATC (n = 480) are assessed before and after training and annually for 5 years on their deployment date; they also complete brief monthly and daily surveys. The RCMP Study results are expected to benefit the mental health of all participants, RCMP and PSP by reducing PTSI among all who serve.

DETAILED DESCRIPTION:
Contemporary programs designed to support PSP mental health focus on increasing knowledge, reducing stigma and increasing help-seeking behaviours. Most studies of PTSI among PSP use cross-sectional data with short follow-up periods and assess very small subsets of variables posited as important. The limited research suggests the extant programs produce small, time-limited, highly variable benefits, likely due to low fidelity of delivery and limited specification of the mechanisms of action for mitigating PTSI. A particularly large, robustly designed trial with serving PSP compared psychoeducation to resilience training focussed on stress reduction and mindfulness, but found no statistically significant differences between the treatment groups. The researchers recommended future programs target specific modifiable individual differences. Individual differences that have been posited as resilience factors for psychopathology include some personality traits (i.e., extroversion, conscientiousness), hope, distress tolerance, optimism, interpersonal supports and positive life activities (e.g., exercise). Environmental factors, individual differences in psychological variables and individual differences in physiological variables have also been posited as risk factors for psychopathology. Environmental risk factors for psychopathology include PPTE and stressors (e.g., adverse childhood experiences, difficult socioeconomic status), family history of psychopathology, pre-existing psychopathology, and peritraumatic experiences. Individual psychological difference risk factors for psychopathology include some personality traits (e.g., neuroticism, world view), anxiety sensitivity, fear of negative evaluation, illness/injury sensitivity, pain-related anxiety/fear, intolerance of uncertainty, rumination, maladaptive self-appraisal, dissociation, and anger. Individual physiological difference risk factors for psychopathology include autonomic nervous system dysregulation. Aversive avoidant reactions to emotions are particularly critical risk factors for developing PTSI. Greater acceptance of emotions reduces reliance on avoidant coping strategies (e.g., alcohol use, avoiding reminders of the event) that exacerbate PTSI symptoms and, paradoxically, lead to more frequent negative emotions. The UP for the transdiagnostic treatment of emotional disorders (UP) is an evidence-based cognitive behaviour intervention designed to help individuals cultivate an approach-oriented stance towards emotions. The UP was designed to reduce symptoms of diverse anxiety- and mood-related disorders. The UP is supported by considerable evidence demonstrating transdiagnostic effectiveness across several delivery formats (e.g., individual, group, self). There is preliminary support for the UP as a proactive intervention to mitigate PTSI based on a randomized trial assessing participants with elevated nonclinical symptoms of depression and anxiety. Participants found the proactive Unified Protocol training to be highly acceptable and satisfying; at 1-month follow-up, they reported using the new skills "some" to "most" of the time, and statistically significant improvements were observed from baseline to 1-month follow-up. The UP appears to have potential as a proactive intervention that can be efficiently and effectively delivered to PSP to use to protect their mental health and enhance job satisfaction.

The RCMP Study necessarily uses a longitudinal prospective sequential experimental cohort design to create a clustered randomized trial that engages individual participants for 5.5 years. The structure of the Cadet Training Program does not allow for randomizing individual participants or individual groups of participants; nevertheless, meta-analytic evidence suggests that results from studies using this design and results from true randomized controlled trials do not typically differ meaningfully or statistically significantly, and both methods produce comparable groups at baseline. The RCMP Study hypotheses were pre-registered with aspredicted.org for the RCMP Study and associated hypotheses occurred on 7 November 2019 with the name, "Risk and resiliency factors in the RCMP: A prospective investigation" (#30654). Participants will be assessed for at least 66 months, via full assessments (i.e., self-report surveys, clinical interviews), monthly assessments (i.e., ~20 minute self-report surveys), daily assessments (i.e., ~1 minute self-report surveys), and biometric assessments, to allow for sufficient time to potentially develop PTSI symptoms after deployment. The data collection time-period uses seven broad milestones (see Table 1 for a summary and the supplemental tables at http://hdl.handle.net/10294/14680 for details): pre-training (T1); pre-deployment (T2; ~26 weeks after recruitment); and each of five deployment anniversaries starting about 12 months after deployment (T3 to T7). Each milestone involves a full assessment (FA1 to FA7). Recruitment will continue until 480 ATC participants have completed FA2. Unless extended by the RCMP, FA7 concludes data collection from each participant. Participants complete their first monthly assessment (i.e., MA1) about 4 weeks after completing FA1 and do not complete a monthly assessment concordant with completion of a full assessment (i.e., maximum number of monthly assessments per participant is 65). Participants can complete their first daily assessment (i.e., DA1) on the same day as FA1 (i.e., maximum number of daily assessments per participant ~2008). Cadets cannot be enrolled into the ATC until all STC participants have deployed, creating a necessarily 26-week gap that will be used to prepare to transition the Cadet Training Program to the ATC (see supplemental tables at http://hdl.handle.net/10294/14680).

1. Mental health disorder prevalence rates at T1 for both groups, based on clinical interviews, or screening tools based on self-reported symptoms, will be comparable to the mental health disorder prevalence rates of the general population (i.e. 10.1%).
2. At T1, both groups will report individual difference scores comparable to the general population.
3. From T1 to T2, both groups will show reductions in variables associated with risk (e.g. anxiety sensitivity), increases in variables associated with resilience (e.g. distress tolerance), improvements in mental health (e.g. absolute, statistically significant or clinically significant reductions in self-reported symptoms of PTSI, reductions in proportions of participants meeting diagnostic criteria using either standardized cut-off scores, clinical interview results), as a function of the Cadet Training Program.

   1. The ATC group will, but the STC participants will not, show statistically significant changes associated with more than small effect sizes.
   2. Relative to the STC group, the ATC group at T2 will report statistically lower risk, greater resilience and better mental health.
4. Both groups will show statistically significant predictive relationships between completing assessments, changes to individual differences over time (i.e. inversely with risk [e.g. anxiety sensitivity], positively with resilience [e.g. hope], inversely with mental health symptoms [e.g. symptoms of major depressive disorder]) and successful completion of the Cadet Training Program.
5. Both groups will evidence statistically significant sequential predictive relationships for environmental factors or individual differences reported during the daily, monthly and full assessments.
6. Both groups will show increases in risk, decreases in resilience and reductions in mental health at T3, T4, T5, T6, and T7, relative to T2; however, the ATC group will show slower increases in risk, slower decreases in resilience and slower reductions in mental health.
7. Both groups will show a statistically significant relationship between changes in environmental factors or individual differences over time, frequency of exercise109 and other self-reported indicators of physical health.
8. Relative to the STC group, the ATC group will report fewer symptoms of and instances of mental health disorders after T1.
9. The ATC group will show a statistically significant relationship between changes in environmental factors or individual differences over time and engagement with ATC content.
10. Relative to men, women will report more difficulties with mental disorder symptoms and occupational stressors.
11. Changes in biological variables (i.e. autonomic nervous system reactivity, heart rate variability, cardiac mechanical changes) will be associated with environmental factors or individual differences.

The RCMP Study has been designed as an applied longitudinal prospective sequential experimental cohort research project. Participants, the RCMP as an organization, past, present and future RCMP and all PSP should benefit directly and indirectly from the RCMP Study. The benefits should occur irrespective of any specific RCMP Study component (i.e. risk variables, resilience variables, biological variables, the relative impact of the ATC). Through the RCMP Study, the RCMP have become global leaders in the international efforts to better support the mental health of all PSP. The current protocol paper provides details to inform and support similar efforts by other researchers.

ELIGIBILITY:
Inclusion Criteria:

* Cadets starting the RCMP Cadet Training Program

Exclusion Criteria:

* Anyone other than cadets starting the RCMP Cadet Training Program

Ages: 19 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 960 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 26) | Time 1 (pre-training; week 1), Time 2 (post-training; week 26)
  Posttraumatic Stress Disorder Checklist Version 5; Total scores range from 0 to 80; Higher scores indicate more severe symptoms.
Sustained Posttraumatic Stress Disorder Symptoms from Time 2 (post-training; week 26) to Time 7 (5-year follow-up) | Time 2 (post-training; week 26), Time 3 (1-year follow-up), Time 4 (2-year follow-up), Time 5 (3-year follow-up), Time 6 (4-year follow-up), Time 7 (5-year follow-up)
  Posttraumatic Stress Disorder Checklist Version 5; Total scores range from 0 to 80; Higher scores indicate more severe symptoms.
Change in Major Depressive Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 26) | Time 1 (pre-training; week 1), Time 2 (post-training; week 26)
  Patient Health Questionnaire - 9 (PHQ-9); Total scores range from 0 to 36; Higher scores indicate more severe symptoms.
Sustained Major Depressive Disorder Symptoms from Time 2 (post-training; week 26) to Time 7 (5-year follow-up) | Time 2 (post-training; week 26), Time 3 (1-year follow-up), Time 4 (2-year follow-up), Time 5 (3-year follow-up), Time 6 (4-year follow-up), Time 7 (5-year follow-up)
  Patient Health Questionnaire - 9 (PHQ-9); Total scores range from 0 to 36; Higher scores indicate more severe symptoms.
Change in Generalized Anxiety Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 26) | Time 1 (pre-training; week 1), Time 2 (post-training; week 26)
  Generalized Anxiety Disorder Scale - 7 (GAD-7); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.
Sustained Generalized Anxiety Disorder Symptoms from Time 2 (post-training; week 26) to Time 7 (5-year follow-up) | Time 2 (post-training; week 26), Time 3 (1-year follow-up), Time 4 (2-year follow-up), Time 5 (3-year follow-up), Time 6 (4-year follow-up), Time 7 (5-year follow-up)
  Generalized Anxiety Disorder Scale - 7 (GAD-7); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.
Change in Panic Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 26) | Time 1 (pre-training; week 1), Time 2 (post-training; week 26)
  Panic Disorder Severity Scale (PDSS); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.
Sustained Panic Disorder Symptoms from Time 2 (post-training; week 26) to Time 7 (5-year follow-up) | Time 2 (post-training; week 26), Time 3 (1-year follow-up), Time 4 (2-year follow-up), Time 5 (3-year follow-up), Time 6 (4-year follow-up), Time 7 (5-year follow-up)
  Panic Disorder Severity Scale (PDSS); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: R. Nicholas Carleton, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
There are ethical and privacy concerns with respect to sharing the participant data, even after anonymization; as such, requests to access the datasets should be directed to the primary investigator and will be addressed on a case-by-case basis in connection with the University of Regina Research Ethics Board.

REFERENCES:
- [Background] Carleton RN, Kratzig GP, Sauer-Zavala S, Neary JP, Lix LM, Fletcher AJ, Afifi TO, Brunet A, Martin R, Hamelin KS, Teckchandani TA, Jamshidi L, Maguire KQ, Gerhard D, McCarron M, Hoeber O, Jones NA, Stewart SH, Keane TM, Sareen J, Dobson K, Asmundson GJG. The Royal Canadian Mounted Police (RCMP) Study: protocol for a prospective investigation of mental health risk and resilience factors. Health Promot Chronic Dis Prev Can. 2022 Aug;42(8):319-333. doi: 10.24095/hpcdp.42.8.02. PMID 35993603
- [Derived] Khoury JMB, Jamshidi L, Shields RE, Nisbet J, Afifi TO, Fletcher AJ, Stewart SH, Asmundson GJG, Sauer-Zavala S, Kratzig GP, Carleton RN. Putative risk and resiliency factors among Royal Canadian Mounted Police cadets. Front Psychol. 2023 Mar 15;14:1048573. doi: 10.3389/fpsyg.2023.1048573. eCollection 2023. PMID 37008880
- See also: RCMP Study Website — https://www.rcmpstudy.ca